CLINICAL TRIAL: NCT02707263
Title: Effect of Intravenous Continuous Infusion Heparin on Rates of Venous Thromboembolism in High-Risk, Critically Ill Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01051
Record Dates: First submitted 2016-03-01; First posted 2016-03-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism
Keywords: heparin
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous continuous infusion of heparin (IV UFH) (Active Comparator): Heparin will be administered intravenously.
  Interventions: Drug: intravenous continuous infusion of heparin (IV UFH)
- Subcutaneous heparin (Active Comparator): Heparin will be subcutaneously administered.
  Interventions: Drug: Subcutaneous Heparin

INTERVENTIONS:
Drug: intravenous continuous infusion of heparin (IV UFH)
  Arms: Intravenous continuous infusion of heparin (IV UFH)
Drug: Subcutaneous Heparin
  Arms: Subcutaneous heparin

SUMMARY:
The primary purpose of this study is to demonstrate that a continuous infusion of intravenous (IV) heparin (UFH) for Venous thromboembolism (VTE) prophylaxis will restore prophylactic levels of heparin in high-risk critically ill medical patients as compared with guideline recommended subcutaneous heparin. Antifactor Xa assay, a laboratory test to measure the anticoagulant activity of heparin, or the ability of heparin to thin the blood, will be used to demonstrate that Intravenous administration is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the medical ICU (MICU)
* High-risk for Venous Thromboembolism (VTE) ≥ 1 of the following:
* Body Mass Index (BMI) ≥ 30 kg/m2
* Personal or family history of VTE
* Receiving vasopressors

Exclusion Criteria:

* Indication for therapeutic anticoagulation
* Evidence of deep vein thrombosis (DVT) on ultrasonography at admission
* Indwelling intrathecal, epidural, or other indwelling deep catheters
* Recent (< 3 months) International Society of Thrombosis and Haemostasis (ISTH) major bleeding13
* Recent (< 3 months) major trauma
* Recent (< 3 months) neurosurgery or orthopedic surgery Pregnancy
* Contraindication to heparin or heparin products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Comparison of Coagulation (Anti-Xa levels) in patients receiving Intravenous Continuous Infusion Heparin versus subcutaneous Heparin | 3 Days

CONTACTS AND LOCATIONS:
Overall Officials: John Papadopoulos, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States